CLINICAL TRIAL: NCT06323161
Title: Efficacy and Safety of Co-administered Cagrilintide and Semaglutide (CagriSema) s.c. in Doses 2.4 mg/2.4 mg and 1.0 mg/1.0 mg Once Weekly Versus Placebo in Participants With Type 2 Diabetes as Add on to Once-daily Basal Insulin With or Without Metformin
Brief Title: A Research Study to See How Much CagriSema Lowers Blood Sugar and Body Weight Compared to Placebo in People With Type 2 Diabetes Treated With Once-daily Basal Insulin With or Without Metformin
Acronym: REIMAGINE 3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9388-7637; U1111-1283-0754 (Other: World Health Organization (WHO)); 2022-502679-43 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CagriSema Dose 1 (Active Comparator): Participants will receive once-weekly subcutaneous (s.c) injections of CagriSema (cagrilintide and semaglutide) at escalating doses every week in 8-week dose escalation period until target dose (dose 1) of CagriSema (cagrilintide and semaglutide) is achieved and maintained up to 32 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- CagriSema Dose 2 (Active Comparator): Participants will receive once-weekly s.c injections of CagriSema (cagrilintide and semaglutide) at escalating doses every week in 16-week dose escalation period until target dose (dose 2) of CagriSema(cagrilintide and semaglutide) is achieved and maintained up to 24 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Placebo Dose 1 (Placebo Comparator): Participants will receive once-weekly s.c injection of placebo matched to cagrisema dose 1 (cagrilintide and semaglutide) for 40 weeks.
  Interventions: Drug: Placebo
- Placebo Dose 2 (Placebo Comparator): Participants will receive once-weekly s.c injection of placebo matched to cagrisema dose 2 (cagrilintide and semaglutide) for 40 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive once-weekly cagrilintide subcutaneously.
  Arms: CagriSema Dose 1; CagriSema Dose 2
Drug: Semaglutide — Participants will receive once-weekly semaglutide subcutaneously.
  Arms: CagriSema Dose 1; CagriSema Dose 2
Drug: Placebo — Participants will receive placebo matched to cagrilintide and semaglutide subcutaneously.
  Arms: Placebo Dose 1; Placebo Dose 2

SUMMARY:
This study will look at how much CagriSema helps people with type 2 diabetes lower their blood sugar and body weight. CagriSema is a new investigational medicine. Doctors may not yet prescribe CagriSema. CagriSema will be compared to a "dummy" medicine (also called "placebo") that has no effect on the body. Participant will get either CagriSema or "dummy" medicine and which treatment they get is decided by chance. Participant will take the study medicine together with their current diabetes medicine (once-daily insulin with or without metformin). For each participant, the study will last for about one year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (sex at birth).
* Age 18 years or above at the time of signing the informed consent.
* Diagnosed with type 2 diabetes mellitus ≥180 days before screening.
* On stable once-daily dose of basal insulin (minimum of 0.25 units per kilogram per day (U/kg/day) or 20 U/day) alone or in combination with metformin (at effective or maximum tolerated dose as judged by the investigator) for 90 days prior to screening.
* Glycated haemoglobin (HbA1c) 7.0-10.5 percent (53-91 millimoles per mole [mmol/mol]) (both inclusive) as determined by central laboratory at screening.
* Body Mass Index (BMI) greater than or equal to 25 kilogram per square meter (kg/m^2) at screening. BMI will be calculated in the electronic case report form (eCRF) based on height and body weight at screening.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using a highly effective contraceptive method.
* Renal impairment with estimated Glomerular Filtration Rate (eGFR) less than 30 milliliters per minute per 1.73 square meter (mL/min/1.73 m^2) as determined by central laboratory at screening.
* Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria within 90 days before screening.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by an eye examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Known hypoglycaemia unawareness as indicated by the investigator according to Clarke's questionnaire question 8.
* Recurrent severe hypoglycaemic episodes within the last year as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-10-23 (Actual)

PRIMARY OUTCOMES:
Change in Glycated Haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 40)
  Measured in percentage (%)- points.

SECONDARY OUTCOMES:
Relative Change in Body Weight | From baseline (week 0) to end of treatment (week 40)
  Measured in percentage (%).
Number of Participants Who Achieve Greater than or Equal to (≥) 10% Body Weight Reduction | From baseline (week 0) to end of treatment (week 40)
  Measured as count of participants.
Number of Participants Who Achieve ≥15% Body Weight Reduction | From baseline (week 0) to end of treatment (week 40)
  Measured as count of participants.
Number of Participants Who Achieve HbA1c Target Values of Less than (<) 7.0% (<53 millimole per mole [mmol/mol]) | At end of treatment (week 40)
  Measured as count of participants.
Number of Participants Who Achieve HbA1c Target Values of Less than or Equal to (≤) 6.5% (≤48 mmol/mol) | At end of treatment (week 40)
  Measured as count of participants.
Change in Fasting Plasma Glucose (FPG) | From baseline (week 0) to end of treatment (week 40)
  Measured as millimole per liter (mmol/L).
Change in Insulin Dose | From baseline (week 0) to end of treatment (week 40)
  Measured in units (u).
Number of Participants Who Achieve Insulin Dose Equal to (=) 0 Units | At end of treatment (week 40)
  Measured as count of participants.
Change in 7-point Self-measured Plasma Glucose (SMPG) Profiles: Mean 7-point profile and Mean postprandial increment (over all meals) | From baseline (week 0) to end of treatment (week 40)
  Measured in mmol/L.
Number of Participants Who Achieve ≥5% Body Weight Reduction | From baseline (week 0) to end of treatment (week 40)
  Measured as count of participants.
Number of Participants Who Achieve ≥20% Body Weight Reduction | From baseline (week 0) to end of treatment (week 40)
  Measured as count of participants.
Change in Waist Circumference | From baseline (week 0) to end of treatment (week 40)
  Measured in centimeter (cm).
Change in Systolic Blood Pressure (SBP) | From baseline (week 0) to end of treatment (week 40)
  Measured in millimeter of mercury (mmHg).
Change in Diastolic Blood Pressure (DBP) | From baseline (week 0) to end of treatment (week 40)
  Measured in mmHg.
Ratio to Baseline in High Sensitivity C-reactive Protein (hsCRP) | From baseline (week 0) to end of treatment (week 40)
  Measured in ratio.
Ratio to Baseline in Lipids: Non-high Density Lipoprotein (Non-HDL) Cholesterol | From baseline (week 0) to end of treatment (week 40)
  Measured in ratio.
Ratio to Baseline in Lipids: Triglycerides | From baseline (week 0) to end of treatment (week 40)
  Measured in ratio.
Ratio to Baseline in Lipids: Low-Density Lipoprotein (LDL) Cholesterol | From baseline (week 0) to end of treatment (week 40)
  Measured in ratio.
Ratio to Baseline in Lipids: Very Low-Density Lipoprotein (VLDL) cholesterol | From baseline (week 0) to end of treatment (week 40)
  Measured in ratio.
Ratio to Baseline in Lipids: HDL Cholesterol | From baseline (week 0) to end of treatment (week 40)
  Measured in ratio.
Ratio to Baseline in Lipids: Total Cholesterol | From baseline (week 0) to end of treatment (week 40)
  Measured in ratio.
Ratio to Baseline in Lipids: Free Fatty Acids | From baseline (week 0) to end of treatment (week 40)
  Measured in ratio.
Change in Short Form-36 Version 2.0 Health Survey (SF-36v2): Vitality score | From baseline (week 0) to end of treatment (week 40)
  Measured as score points. SF-36v2 Acute measures Health-Related Quality of Life (HRQoL). The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 Acute scores are norm-based scores, that is. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Higher scores indicate better functional health and well-being. The vitality score range is from 25.6 to 69.1.
Change in SF-36v2: Physical Component Summary Score | From baseline (week 0) to end of treatment (week 40)
  Measured as score points. SF-36v2 Acute measures HRQoL. The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 Acute scores are norm-based scores, that is. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Higher scores indicate better functional health and well-being. The score range for physical component summary is 6.1 to 79.7.
Change in SF-36v2: Mental Component Summary Core | From baseline (week 0) to end of treatment (week 40)
  Measured as score points. SF-36v2 Acute measures HRQoL. The measure consists of 36 items yielding 8 health domain scores and 2 component summary scores. SF-36v2 Acute scores are norm-based scores, that is. transformed to a scale where the 2009 US general population has a mean of 50 and a standard deviation of 10. Higher scores indicate better functional health and well-being. The score range for mental component summary score is -3.8 to 78.7.
Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ) Score | From baseline (week 0) to end of treatment (week 40)
  Measured as score points. DTSQs measures treatment satisfaction and diabetes-specific quality of life. The measure consists of 8 items yielding 1 global score and 2 single item scores. Higher scores on the global score indicate greater satisfaction with treatment. Lower scores on the single-item scores indicate BG levels closer to the ideal, while higher scores indicate problems. Single-item scores (score range): Perceived frequency of hyperglycaemia (0-6), Perceived frequency of hypoglycaemia (0-6). Global score (score range): Total Treatment Satisfaction (0-36).
Ratio to Baseline in Leptin | From baseline (week 0) to end of treatment (week 40)
  Measured in ratio.
Ratio to Baseline in Soluble Leptin Receptor | From baseline (week 0) to end of treatment (week 40)
  Measured in ratio.
Number of Treatment Emergent Adverse Events (TEAEs) | From baseline (week 0) to end of treatment +7 weeks (week 47)
  Measured as count of events.
Number of Clinically Significant Hypoglycaemic Episodes (level 2) (<3.0 mmol/L (54 mg/dL), Confirmed by Blood Glucose Meter) | From baseline (week 0) to end of treatment +7 weeks (week 47)
  Measured as count of episodes.
Number of Clinically Significant Hypoglycaemic Episodes (level 3) | From baseline (week 0) to end of treatment +7 weeks (week 47)
  Measured as count of episodes. Hypoglycaemic episodes (level 3) is hypoglycaemia associated with severe cognitive impairment requiring external assistance for recovery, with no specific glucose threshold.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (53):
- United States (14):
  - Valley Clinical Trials, Inc., Northridge, California
  - Bioclinical Research Alliance, Miami, Florida
  - Solaris Clinical Research, Meridian, Idaho
  - Iowa Diab & Endo Res Center, West Des Moines, Iowa
  - Alliance for Multispec Res, Newton, Kansas
  - Elite Research Center, Flint, Michigan
  - Palm Research Center Inc., Las Vegas, Nevada
  - University of North Carolina, Chapel Hill, North Carolina
  - Clinical Research Associates, Nashville, Tennessee
  - Velocity Clinical Res-Dallas, Dallas, Texas
  - Synergy Groups Medical, Houston, Texas
  - PlanIt Research, PLLC, Houston, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - TPMG Clinical Research, Newport News, Virginia
- China (9):
  - Chinese People's Liberation Army General Hospital-Endocrinology, Beijing, Beijing Municipality
  - Huaihe Hospital of Henan University-Endocrinology, Kaifeng, Henan
  - Huaihe Hospital of Henan University, Kaifeng, Henan
  - The Second Affiliated Hospital of Nanjing Medical University-Endocrinology, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University_Nanjing, Nanjing, Jiangsu
  - The Affiliated Hospital of Jiangsu University-Endocrinology, Zhenjiang, Jiangsu
  - Jinan Central Hospital, Ji'nan, Shandong
  - Jinan Central Hospital Affiliated to Shandong University, Jinan, Shandong
  - Shanghai Pudong New Area People's Hospital-Endocrinology, Shanghai, Shanghai Municipality
- Japan (15):
  - Manda Memorial Hospital_Internal Medicine, Sapporo-shi, Hokkaido, Hokkaido, Japan
  - Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi, Kanagawa
  - Kumanomae Nishimura Naika Clinic_Internal Medicine, Arakawa-ku, Tokyo
  - Akaicho Clinic, Chiba-shi, Chiba
  - Futata Tetsuhiro Clinic Meinohama_Internal medicine, Fukuoka-shi, Fukuoka
  - Kunisaki Makoto Clinic, Fukuoka-shi, Fukuoka
  - Sasaki Internal Medicine, Hokkaido
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - H.E.C Science Clinic, Kanagawa
  - Kyoto University Hospital, Kyoto-shi, Kyoto
  - Minami Akatsuka Clinic, Mito-shi, Ibaraki
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Tokyo-Eki Center-building Clinic, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Kato Clinic of Internal Medicine_Internal Medicine, Tokyo
- Serbia (5):
  - Healthcare centre Zvezdara, Belgrade, RS
  - Healthcare centre Kragujevac, Kragujevac, RS
  - University Clinical Centre Nis, Niš, RS
  - Healthcare centre Nis, Niš, RS
  - Policlinic for diabetes, Zaječar
- Slovakia (5):
  - MOMED, s.r.o, Kráľovský Chlmec
  - DIA - KONTROL s.r.o., Levice
  - SIN AZUCAR s.r.o., Malacky
  - ENRIN, s.r.o., Rimavská Sobota
  - LUDIA, s. r. o., Spišská Nová Ves
- South Africa (5):
  - Oraderumaz (Pty) Ltd, Bloemfontein, Free State
  - Lenasia Clinical Trial Centre, Lenasia, Gauteng
  - Prinshof Medical Campus, Pretoria, Gauteng
  - Clinical Trial Systems (CTC), Pretoria, Gauteng
  - Ashmed Medi-Centre, Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com